CLINICAL TRIAL: NCT00756600
Title: A Multi-site Randomised Controlled Trial Comparing Regional and General Anaesthesia for Effects on Neurodevelopmental Outcome and Apnoea in Infants
Brief Title: A Multi-site Randomized Controlled Trial Comparing Regional and General Anesthesia for Effects on Neurodevelopmental Outcome and Apnea in Infants
Acronym: GAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Royal Children's Hospital (Other); Royal Hospital for Sick Children (Other); Murdoch Childrens Research Institute (Other); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mary Ellen McCann, MD, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06-07-0320
Record Dates: First submitted 2008-09-18; First posted 2008-09-22 (Estimated); Results first posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Inguinal Hernia
Keywords: Infants; scheduled; unilateral; bilateral; repair
MeSH Terms: conditions — Hernia, Inguinal | interventions — Anesthesia, Conduction; Anesthesia, Spinal; Anesthesia, General

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 1 (Active Comparator): Regional Anesthesia
  Interventions: Drug: Regional Anesthesia
- 2 (Active Comparator): General Anesthesia
  Interventions: Drug: General Anesthesia

INTERVENTIONS:
Drug: Regional Anesthesia — Up to 2.5 mg/kg bupivacaine administered by caudal or subarachnoid routes or both caudal and subarachnoid or subarachnoid and ilioinguinal nerve blockade. Single shot.
  Other Names: Spinal Anesthesia.
  Arms: 1
Drug: General Anesthesia — Sevoflurane for induction and maintenance of general anesthesia, dose up to 8% inspired for duration of procedure plus bupivacaine local anesthetic blockade (up to 2.5 mg/kg) administered via caudal or ilioinguinal nerve block.
  Other Names: General Anesthesia.
  Arms: 2

SUMMARY:
The primary purpose of the GAS study is to determine whether different types of anesthesia (Regional versus General) given to 720 infants undergoing inguinal hernia repair results in equivalent neurodevelopmental outcomes. The study also aims to describe the incidence of apnea in the post-operative period after both regional and general anesthesia for inguinal hernia repair in infants. This study is important as it will provide the greatest evidence for safety or toxicity of general anesthesia for human infants.

DETAILED DESCRIPTION:
This is a prospective, observer blind, multi-site, randomized, controlled, equivalence trial. The general anesthesia group will receive sevoflurane (intervention drug) for induction and maintenance of general anesthesia, dose up to 8% inspired for duration of procedure plus bupivacaine local anesthetic blockade (up to 2.5 mg per kg) administered via caudal or ilioinguinal nerve block. The airway can be maintained with a face mask, laryngeal mask or endotracheal tube, with or without neuromuscular blocking agents.

The regional group will have no sedative agent. The regional blockade may be with spinal alone, spinal block with caudal block, spinal with ilioinguinal block or caudal alone. The maximum dose of 2.5 mg per kg of bupivacaine can be used.

ELIGIBILITY:
Inclusion Criteria:

* Any infant scheduled for unilateral or bilateral inguinal hernia repair (with or without circumcision)
* Any infant whose gestational age is 26 weeks or more (GA = 182 days)
* Any infant whose post-menstrual age is up to 60 weeks (PMA = 426 days)

Exclusion Criteria:

* Any child older than 60 weeks post-menstrual age
* Any child born less than 26 weeks gestation
* Any contraindication to general or spinal/caudal anesthesia (for example: neuromuscular disorder or coagulopathy)
* Pre-operative ventilation immediately prior to surgery
* Congenital heart disease that has required ongoing pharmacotherapy
* Known chromosomal abnormality or any other known acquired or congenital abnormalities (apart from prematurity) which are likely to affect development
* Children where follow-up would be difficult for geographic or social reasons
* Families where English is not the primary language spoken at home
* Known neurological injury such as cystic periventricular leukomalacia (PVL), or grade 3 or 4 intra ventricular hemorrhage (ICH) (+/- post hemorrhage ventricular dilation)
* Previous exposure to volatile anesthesia or benzodiazepines as a neonate or in the third trimester in utero.

Max Age: 60 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 643 (Actual)
Dates: Start 2006-10-23 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Davidson, MD, Principal Investigator — Royal Children's Hospital, Victoria, Australia; Mary Ellen McCann, MD, Principal Investigator — Children's Hospital Boston, United States of America; Neil Morton, MD, Principal Investigator — Royal Hospital for Sick Children, Glasgow, United Kingdom
Locations (30):
- United States (10):
  - The Children's Hospital Denver, Aurora, Colorado
  - Children's Memorial Hospital, Chicago, Illinois
  - The University of Iowa Hospital, Iowa City, Iowa
  - Children's Hospital Boston, Boston, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Children's Medical Center of Dallas, Dallas, Texas
  - Vermont Children's Hospital at Fletcher Allen Health Care, Burlington, Vermont
  - Seattle Children's Hospital, Seattle, Washington
- Australia (6):
  - Adelaide Women's and Children's Hospital, North Adelaide, South Australia
  - Casey Hospital, Berwick, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Cabrini Hospital, Malvern, Victoria
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital, Perth, Western Australia
- Canada (2):
  - Montreal Children's Hospital, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
- Italy (3):
  - Ospedali Riuniti Di Bergamo, Bergamo
  - G. Gaslini Children's Hospital, Genoa
  - 'Vitore Buzzi' Children's Hospital, Milan
- Netherlands (2):
  - Universitair Medisch Centrum Groningen, Groningen
  - Wilhelmina Children's Hospital; University Medical Centre Utrecht, Utrecht
- Starship Children's Health, Auckland, New Zealand
- United Kingdom (6):
  - Royal Belfast Hospital for Sick Children, Belfast
  - Birmingham Children's Hospital, Birmingham
  - Bristol Royal Hospital for Children, Bristol
  - Royal Hospital for Sick Children, Glasgow
  - Royal Liverpool Children's Hospital, Liverpool
  - Sheffield Children's Hospital, Sheffield

REFERENCES:
- [Background] Davidson A, McCann ME, Morton N. Anesthesia neurotoxicity in neonates: the need for clinical research. Anesth Analg. 2007 Sep;105(3):881-2. doi: 10.1213/01.ane.0000269692.57331.48. No abstract available. PMID 17717261
- [Derived] McCann ME, de Graaff JC, Dorris L, Disma N, Withington D, Bell G, Grobler A, Stargatt R, Hunt RW, Sheppard SJ, Marmor J, Giribaldi G, Bellinger DC, Hartmann PL, Hardy P, Frawley G, Izzo F, von Ungern Sternberg BS, Lynn A, Wilton N, Mueller M, Polaner DM, Absalom AR, Szmuk P, Morton N, Berde C, Soriano S, Davidson AJ; GAS Consortium. Neurodevelopmental outcome at 5 years of age after general anaesthesia or awake-regional anaesthesia in infancy (GAS): an international, multicentre, randomised, controlled equivalence trial. Lancet. 2019 Feb 16;393(10172):664-677. doi: 10.1016/S0140-6736(18)32485-1. Epub 2019 Feb 14. PMID 30782342
- [Derived] Davidson AJ, Disma N, de Graaff JC, Withington DE, Dorris L, Bell G, Stargatt R, Bellinger DC, Schuster T, Arnup SJ, Hardy P, Hunt RW, Takagi MJ, Giribaldi G, Hartmann PL, Salvo I, Morton NS, von Ungern Sternberg BS, Locatelli BG, Wilton N, Lynn A, Thomas JJ, Polaner D, Bagshaw O, Szmuk P, Absalom AR, Frawley G, Berde C, Ormond GD, Marmor J, McCann ME; GAS consortium. Neurodevelopmental outcome at 2 years of age after general anaesthesia and awake-regional anaesthesia in infancy (GAS): an international multicentre, randomised controlled trial. Lancet. 2016 Jan 16;387(10015):239-50. doi: 10.1016/S0140-6736(15)00608-X. Epub 2015 Nov 4. PMID 26507180

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There are no significant events that occur after enrollment and before randomization.
Period: Overall Study
Arm/Group | Regional Anesthesia | General Anesthesia
Started | 287 | 356
Completed | 287 | 356
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Not all patients returned for their follow up visit. For this reason, only 205 participants in the "Regional Anesthesia" group and 242 participants in the "General Anesthesia" group were included in the published analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Regional Anesthesia | General Anesthesia | Total
Number analyzed (Participants) | 287 | 356 | 643
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 287 | 356 | 643
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: days] | 68.9 (30.8) | 71.1 (31.7) | 70 (NA) — Data required to calculate the total standard deviation could not be found despite all efforts to locate the underlying data
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 52 | 107
  Male | 232 | 304 | 536
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Population: Not all patients returned for their follow up visit. For this reason, only 205 participants in the "Regional Anesthesia" group and 242 participants in the "General Anesthesia" group total were included in the published analysis.
  The number of participants from each region were the only ones ultimately analyzed and published.
  participants
    New Zealand: number analyzed (Participants) | 205 | 242 | 447
    New Zealand | 7 | 9 | 16
    Canada: number analyzed (Participants) | 205 | 242 | 447
    Canada | 10 | 20 | 30
    Netherlands: number analyzed (Participants) | 205 | 242 | 447
    Netherlands | 19 | 17 | 36
    United States: number analyzed (Participants) | 205 | 242 | 447
    United States | 34 | 52 | 86
    Italy: number analyzed (Participants) | 205 | 242 | 447
    Italy | 45 | 50 | 95
    United Kingdom: number analyzed (Participants) | 205 | 242 | 447
    United Kingdom | 27 | 22 | 49
    Australia: number analyzed (Participants) | 205 | 242 | 447
    Australia | 63 | 72 | 135

OUTCOME MEASURES:

1. Primary Outcome: Full Scale IQ Score
Description: The primary outcome will be the Wechsler Preschool and Primary Scale of Intelligence-Third Edition (WPPSI-III) full scale IQ score. Verbal, visuo-spatial and processing speed skills are incorporated into the Full Scale IQ score, which is indicative of general intellectual ability.
  Minimum score: 45 Maximum score:145 Higher scores are associated with higher IQ scores (better outcome).
  Note: Scale ranges represent estimates that are very likely to be accurate but which will be verified after access to the physical assessment booklets is restored. The current health situation prohibits the research team from verifying this information at the moment.
Time Frame: At 5 years chronological age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 205 | 242
score on scale | 100.5 (14.3) | 100.1 (15.3)

2. Secondary Outcome: Verbal IQ
Description: Wechsler Preschool and Primary Scale of Intelligence, Third Edition (WPPSI-III): Verbal IQ
  Minimum possible score:45 Maximum possible score:145
  A higher score indicates higher verbal IQ (better outcome).
  Note: Scale ranges represent estimates that are very likely to be accurate but which will be verified after access to the physical assessment booklets is restored. The current health situation prohibits the research team from verifying this information at the moment.
Time Frame: At 5 years corrected age.
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 206 | 240
score on scale | 101.8 (14.7) | 100.9 (15.4)

3. Secondary Outcome: Performance IQ
Description: Wechsler Preschool and Primary Scale of Intelligence, Third Edition (WPPSI-III): Performance IQ
  Minimum possible score:45 Maximum possible score:145
  A higher score indicates a higher performance IQ (better outcome).
  Note: Scale ranges represent estimates that are very likely to be accurate but which will be verified after access to the physical assessment booklets is restored. The current health situation prohibits the research team from verifying this information at the moment.
Time Frame: At 5 years corrected age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 206 | 241
score on scale | 100.7 (15.2) | 101.2 (15.9)

4. Secondary Outcome: Processing Speed Quotient
Description: Wechsler Preschool and Primary Scale of Intelligence, Third Edition (WPPSI-III): Processing speed quotient
  Minimum possible score:45 Maximum possible score:145
  A higher score indicates a better outcome.
  Note: Scale ranges represent estimates that are very likely to be accurate but which will be verified after access to the physical assessment booklets is restored. The current health situation prohibits the research team from verifying this information at the moment.
Time Frame: At 5 years corrected age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 196 | 220
score on scale | 95.8 (14.5) | 96.3 (15.4)

5. Secondary Outcome: Sentence Repetition Scaled Score
Description: Developmental Neuropsychological Assessment second edition (NEPSY-II) sub test: Sentence Repetition scaled score
  Minimum possible score: 1 Maximum possible score: 19
  A higher score indicates a better outcome.
Time Frame: At 5 years chronological age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 175 | 202
score on scale | 9.7 (2.9) | 9.7 (2.8)

6. Secondary Outcome: Auditory Attention Combined Scaled Score
Description: Developmental Neuropsychological Assessment Second Edition (NEPSY-II) Sub Test: Auditory Attention combined scaled score
  Minimum possible score: 1 Maximum possible score: 19
  A higher score indicates a better outcome.
Time Frame: At 5 years corrected age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 167 | 183
score on scale | 9.0 (2.7) | 9.3 (3.0)

7. Secondary Outcome: Statue Scaled Score
Description: Developmental Neuropsychological Assessment Second Edition (NEPSY-II) Sub Test: Statue scaled score
  Minimum possible score: 1 Maximum possible score: 19
  A higher score indicates a better outcome.
Time Frame: At 5 years corrected age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 160 | 182
score on scale | 8.8 (3.5) | 8.6 (3.6)

8. Secondary Outcome: Inhibition Combined Scaled Score
Description: Developmental Neuropsychological Assessment Second Edition (NEPSY-II) Sub Test: Inhibition combined scaled score
  Minimum possible score: 1 Maximum possible score: 19
  A higher score indicates a better outcome.
Time Frame: At 5 years corrected age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 150 | 160
score on scale | 8.3 (3.1) | 8.9 (3.0)

9. Secondary Outcome: Word Generation Scaled Score
Description: Developmental Neuropsychological Assessment Second Edition (NEPSY-II) Sub Test: Word Generation Scaled score
  Minimum possible score: 1 Maximum possible score: 19
  A higher score indicates a better outcome.
Time Frame: At 5 years corrected age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 182 | 199
score on scale | 9.4 (3.4) | 9.3 (3.3)

10. Secondary Outcome: Affect Recognition Scaled Score
Description: Developmental Neuropsychological Assessment Second Edition (NEPSY-II) Sub Test: Affect Recognition scaled score
  Minimum possible score: 1 Maximum possible score: 19
  A higher score indicates a better outcome.
Time Frame: At 5 years corrected age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 174 | 208
score on scale | 10.6 (2.8) | 10.4 (3.2)

11. Secondary Outcome: Memory for Names and Memory for Names Delay
Description: Developmental Neuropsychological Assessment Second Edition (NEPSY-II) Sub Test: Memory for Names and Memory for Names Delay
  Minimum possible score: 1 Maximum possible score: 19
  A higher score indicates a better outcome.
Time Frame: At 5 years corrected age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 180 | 208
score on scale | 8.1 (3.2) | 8.1 (3.2)

12. Secondary Outcome: Theory of Mind Scaled Score
Description: Developmental Neuropsychological Assessment Second Edition (NEPSY-II) Sub Test: Theory of Mind scaled score
  Minimum possible score: 1 Maximum possible score: 19
  A higher score indicates a better outcome.
Time Frame: At 5 years corrected age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 163 | 178
score on scale | 9.8 (2.9) | 9.3 (3.0)

13. Secondary Outcome: Speeded Naming Combined Scaled Score
Description: Developmental Neuropsychological Assessment Second Edition (NEPSY-II) Sub Test: Speeded Naming combined scaled score
  Minimum possible score: 1 Maximum possible score: 19
  A higher score indicates a better outcome.
Time Frame: At 5 years corrected age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Mean (Standard Deviation); unit: score on scale
Groups:
- Regional Anesthesia1: Regional Anesthesia: Up to 2.5 mg/kg bupivacaine administered by caudal or subarachnoid routes or both caudal and subarachnoid or subarachnoid and ilioinguinal nerve blockade. Single shot.
Arm/Group | Regional Anesthesia1 | General Anesthesia
Number analyzed (Participants) | 132 | 142
score on scale | 9.7 (3.0) | 9.8 (3.2)

14. Secondary Outcome: Fingertip Tapping Repetitions Scaled Score
Description: Developmental Neuropsychological Assessment Second Edition (NEPSY-II) Sub Test:Fingertip tapping repetitions scaled score
  Minimum possible score: 1 Maximum possible score: 19
  A higher score is indicative of a better outcome.
Time Frame: At 5 years corrected age
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 180 | 195
score on scale | 9.8 (3.4) | 9.7 (3.4)

15. Secondary Outcome: Fingertip Tapping Sequences Scaled Score
Description: Developmental Neuropsychological Assessment Second Edition (NEPSY-II) Sub Test: fingertip tapping sequences scaled score
  Minimum possible score: 1 Maximum possible score: 19
  A higher score indicates a better outcome.
Time Frame: At 5 years corrected age
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 173 | 183
score on scale | 8.1 (3.4) | 7.7 (3.6)

16. Secondary Outcome: Design Copy Process Total Scaled Score
Description: Developmental Neuropsychological Assessment Second Edition (NEPSY-II) Sub Test: Design Copy Process Total Scaled Score
  Minimum possible score: 1 Maximum possible score: 19
  A higher score indicates a better outcome.
Time Frame: At 5 years corrected age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 172 | 207
score on a scale | 9.6 (3.4) | 9.9 (3.1)

17. Secondary Outcome: Word Reading Standard Score
Description: Weschler Individual Achievement Test (WIAT-II Abbreviated) to assess the academic skills of the child: Word Reading standard score
  Minimum possible score: 45 Maximum possible score: 145
  Note: Scale ranges represent estimates that are very likely to be accurate but which will be verified after access to the physical assessment booklets is restored. The current health situation prohibits the research team from verifying this information at the moment.
  A higher score indicates a better outcome.
Time Frame: At 5 years chronological age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 147 | 167
score on scale | 92.3 (18.1) | 92.8 (211)

18. Secondary Outcome: Numerical Operations Standard Score
Description: Weschler Individual Achievement Test (WIAT-II Abbreviated) to Assess the Academic Skills of the Child: Numerical Operations standard score
  Minimum possible score: 45 Maximum possible score: 145
  Note: Scale ranges represent estimates that are very likely to be accurate but which will be verified after access to the physical assessment booklets is restored. The current health situation prohibits the research team from verifying this information at the moment.
  A higher score indicates a better outcome.
Time Frame: At 5 years chronological age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 146 | 161
score on scale | 98.8 (16.2) | 96.2 (20.8)

19. Secondary Outcome: Spelling Standard Score
Description: Weschler Individual Achievement Test (WIAT-II Abbreviated) to Assess the Academic Skills of the Child: Spelling standard score
  Minimum possible score: 45 Maximum possible score: 145
  A higher score indicates a better outcome.
  Note: Scale ranges represent estimates that are very likely to be accurate but which will be verified after access to the physical assessment booklets is restored. The current health situation prohibits the research team from verifying this information at the moment.
Time Frame: At 5 years chronological age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 141 | 152
score on scale | 90.1 (13.2) | 90.8 (16.5)

20. Secondary Outcome: Numbers Total Scaled Score
Description: Children's Memory Scale (CMS):Numbers Total scaled score
  Minimum possible score: 1 Maximum possible score: 19
  A higher score indicates a better outcome.
Time Frame: At 5 years chronological age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 194 | 229
score on scale | 8.3 (3.2) | 8.1 (3.4)

21. Secondary Outcome: Word Lists 1 (Learning) Scaled Score
Description: Children's Memory Scale (CMS): Word Lists 1 (learning) scaled score
  Minimum possible score: 1 Maximum possible score: 19
  A higher score indicates a better outcome.
Time Frame: At 5 years chronological age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 186 | 224
score on scale | 8.3 (3.4) | 8.6 (3.5)

22. Secondary Outcome: Memory and Learning Word Lists II (Delayed) Scaled Score
Description: Children's Memory Scale (CMS): Memory and learning Word Lists II (delayed) scaled score
  Minimum possible score: 1 Maximum possible score: 19
  A higher score indicates a better outcome.
Time Frame: At 5 years chronological age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 178 | 209
score on scale | 9.7 (2.8) | 9.6 (2.9)

23. Secondary Outcome: The Global Executive Composite (GEC) of the Behaviour Rating of Executive Function
Description: Full title: The Global Executive Composite (GEC) of the Behaviour Rating of Executive Function
  Preschool Version Parent Form (BRIEF-P) to measure behavioural executive abilities.
  Minimum possible score: 40 Maximum possible score: 110
  Note: Scale ranges represent estimates that are very likely to be accurate but which will be verified after access to the physical assessment booklets is restored. The current health situation prohibits the research team from verifying this information at the moment.
  A higher score indicates a worse outcome.
Time Frame: At 5 years chronological age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 198 | 232
score on scale | 48.4 (12.5) | 51.5 (13.4)

24. Secondary Outcome: The Global Adaptive Composite (GAC) of the Adaptive Behavior Assessment System
Description: Full title: The Global Adaptive Composite (GAC) of the Adaptive Behavior Assessment System
  - 2nd edition (ABAS-II) to measure the child's adaptive behavior.
  Minimum possible score: 45 Maximum possible score: 145
  A higher score indicates a better outcome.
  Note: Scale ranges represent estimates that are very likely to be accurate but which will be verified after access to the physical assessment booklets is restored. The current health situation prohibits the research team from verifying this information at the moment.
Time Frame: At 5 years chronological age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 168 | 200
score on scale | 95.9 (16.3) | 94.1 (16.5)

25. Secondary Outcome: Total Problems Score
Description: Child Behaviour Checklist Caregiver Questionnaire (CBCL): Total Problems Score to measure behavioural problems
  Minimum possible score: 40 Maximum possible score: 100
  A higher score indicates a worse outcome.
  Note: Scale ranges represent estimates that are very likely to be accurate but which will be verified after access to the physical assessment booklets is restored. The current health situation prohibits the research team from verifying this information at the moment.
Time Frame: At 5 years chronological age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 215 | 254
score on scale | 44.6 (11.7) | 46.7 (12.5)

26. Secondary Outcome: Internalising Problems T Score
Description: Child Behaviour Checklist Caregiver Questionnaire (CBCL): CBCL internalising problems T score
  Minimum possible score: 40 Maximum possible score: 100
  A higher score indicates a worse outcome.
  Note: Scale ranges represent estimates that are very likely to be accurate but which will be verified after access to the physical assessment booklets is restored. The current health situation prohibits the research team from verifying this information at the moment.
Time Frame: At 5 years chronological age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 215 | 254
score on scale | 46.1 (12.5) | 48.0 (12.5)

27. Secondary Outcome: Externalising Problems T Score
Description: Child Behaviour Checklist Caregiver Questionnaire (CBCL): externalising problems T score
  Minimum possible score: 40 Maximum possible score: 100
  A higher score indicates a worse outcome.
  Note: Scale ranges represent estimates that are very likely to be accurate but which will be verified after access to the physical assessment booklets is restored. The current health situation prohibits the research team from verifying this information at the moment.
Time Frame: At 5 years chronological age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 215 | 254
score on scale | 44.0 (10.7) | 45.8 (11.9)

28. Secondary Outcome: Speech or Language Interventions
Description: Speech or language issues/interventions. These variables will be summarised using descriptive statistics by treatment arm only. No treatment effect or confidence intervals will be calculated.
Time Frame: At 5 years chronological age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Number; unit: participants
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 214 | 257
participants | 18 | 17

29. Secondary Outcome: Psychomotor Interventions
Description: Psychomotor issues/interventions. These variables will be summarised using descriptive statistics by treatment arm only. No treatment effect or confidence intervals will be calculated.
Time Frame: At 5 years chronological age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Number; unit: participants
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 214 | 257
participants | 8 | 6

30. Secondary Outcome: Number of Participants With Global Developmental Delay
Description: Child has global developmental delay. These variables will be summarised using descriptive statistics by treatment arm only. No treatment effect or confidence intervals will be calculated.
Time Frame: At 5 years chronological age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Number; unit: participants
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 204 | 238
participants | 2 | 0

31. Secondary Outcome: Number of Participants With Attention Deficit Hyperactivity Disorder
Description: Child has been diagnosed with Attention Deficit Hyperactivity Disorder. These variables will be summarised using descriptive statistics by treatment arm only. No treatment effect or confidence intervals will be calculated.
Time Frame: At 5 years chronological age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Number; unit: participants
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 214 | 257
participants | 3 | 4

32. Secondary Outcome: Number of Participants With Autism Spectrum Disorder
Description: Child has been diagnosis with Autism Spectrum Disorder. These variables will be summarised using descriptive statistics by treatment arm only. No treatment effect or confidence intervals will be calculated.
Time Frame: At 5 years chronological age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Number; unit: participants
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 211 | 251
participants | 5 | 11

33. Secondary Outcome: Number of Participants With a Hearing Abnormality
Description: Child has a hearing abnormality. These variables will be summarised using descriptive statistics by treatment arm only. No treatment effect or confidence intervals will be calculated.
Time Frame: At 5 years chronological age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Number; unit: participants
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 213 | 252
participants | 8 | 11

34. Secondary Outcome: Number of Participants With a Visual Defect in Either Eye
Description: Child has a visual defect in either eye. These variables will be summarised using descriptive statistics by treatment arm only. No treatment effect or confidence intervals will be calculated.
Time Frame: At 5 years chronological age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Number; unit: participants
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 213 | 254
participants | 21 | 31

35. Secondary Outcome: Number of Participants With a Hearing Aid
Description: Child has a hearing aid. These variables will be summarised using descriptive statistics by treatment arm only. No treatment effect or confidence intervals will be calculated.
Time Frame: At 5 years chronological age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Number; unit: participants
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 211 | 251
participants | 0 | 3

36. Secondary Outcome: Number of Participants Who Are Legally Blind
Description: Child is legally blind. These variables will be summarised using descriptive statistics by treatment arm only. No treatment effect or confidence intervals will be calculated.
Time Frame: At 5 years chronological age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Number; unit: participants
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 212 | 254
participants | 0 | 0

37. Secondary Outcome: Number of Participants Who Have Cerebral Palsy
Description: Child has cerebral palsy. These variables will be summarised using descriptive statistics by treatment arm only. No treatment effect or confidence intervals will be calculated.
Time Frame: At 5 years chronological age
Population: Not all participants had data collected for this Outcome Measure due to absence at follow up visit.
Measure: Number; unit: participants
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 213 | 254
participants | 1 | 3

38. Secondary Outcome: Parents' Awareness of Group Allocation
Description: Whether or not a parent is aware of which treatment group their child was allocated to. This variable will be summarised using descriptive statistics by treatment arm only. No treatment effect or confidence intervals will be calculated.
Time Frame: At 5 years chronological age
Measure: Number; unit: caregivers
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 287 | 356
caregivers | 105 | 118

39. Secondary Outcome: Awareness of Group Allocation by Psychologist
Description: These variables will be summarised using descriptive statistics by treatment arm only. No treatment effect or confidence intervals will be calculated.
Time Frame: At 5 years chronological age
Measure: Number; unit: psychologists
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 287 | 356
psychologists | 7 | 7

40. Secondary Outcome: Awareness of Group Allocation by Pediatrician
Time Frame: At 5 years chronological age
Measure: Number; unit: Pediatricians
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 287 | 356
Pediatricians | 13 | 13

ADVERSE EVENTS:
Time Frame: Adverse Events were not monitored/assessed
Description: Adverse Events were not monitored/assessed
Arm/Group | Regional Anesthesia | General Anesthesia
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-27): https://cdn.clinicaltrials.gov/large-docs/00/NCT00756600/Prot_SAP_000.pdf